CLINICAL TRIAL: NCT00704678
Title: A 12-week, Open Label, Multicenter, Titration Study, With a 12 Month Extension, to Determine the Optimal Titration Regimen for SBR759, Compared to Sevelamer HCl, in Lowering Serum Phosphate Levels in Asian Patients With Chronic Kidney Disease on Hemodialysis
Brief Title: Optimal Titration Regimen for SBR759 in Lowering Serum Phosphate Levels in Asian Chronic Kidney Disease Patients on Hemodialysis
Acronym: SBR759
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSBR759A2202
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; hemodialysis; hyperphosphatemia; Asian; patients
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia | interventions — SBR 759; Sevelamer

ARMS (4):
- 1 (Experimental): 1g bid
  Interventions: Drug: SBR759
- 2 (Active Comparator): 0.8 g tid
  Interventions: Drug: Sevelamer HCl
- 3 (Experimental): 1.5 g tid
  Interventions: Drug: Sevelamer HCl
- 4 (Active Comparator): 1.6 g tid
  Interventions: Drug: Sevelamer HCl

INTERVENTIONS:
Drug: SBR759 — 1g tid
  Arms: 1
Drug: Sevelamer HCl — 1.6 g tid
  Arms: 4
Drug: Sevelamer HCl — 1.5 g tid
  Arms: 3
Drug: Sevelamer HCl — 0.8 g tid
  Arms: 2

SUMMARY:
This study will determine the titration regimen for SBR759 compared to sevelamer HCl in lowering serum phosphate levels in Asian Chronic Kidney Disease patients on hemodialysis

ELIGIBILITY:
Inclusion criteria

* Men or women of at least 18 years old or 20 years old in Japan.
* Stable maintenance of hemodialysis 3 times per week.
* Controlled serum phosphate if under phosphate-binder therapy.
* Serum phosphate level > 6.0 mg/dL (> 1.9 mmol/L) prior to study treatment initiation.

Exclusion criteria

* Peritoneal dialysis or a non-conventional hemodialysis technique .
* Parathyroidectomy or transplant scheduled during the study.
* Uncontrolled hyperparathyroidism
* History of hemochromatosis or ferritin > 800 µg/L.
* Clinically significant GI disorder
* Unstable medical condition other than Chronic Kidney Disease.
* Treated with sevelamer HCl monotherapy or SBR759.
* Treated with oral iron.
* Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2008-08; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Responder rates achieving target serum phosphate levels. | Week 12

SECONDARY OUTCOMES:
Responder rates in target patients with serum calcium-phosphate levels. | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (15):
- Japan (12):
  - Novartis Investigative Site, Kōriyama, Fukushima
  - Novartis Investigative Site, Midori, Gunma
  - Novartis Investigative Site, Hitachiomiya, Ibaraki
  - Novartis Investigative Site, Moriya, Ibaraki
  - Novartis Investigative Site, Sashima-gun, Ibaraki
  - Novartis Investigative Site, Takamatsu, Kagawa-ken
  - Novartis Investigative Site, Tsu, Mie-ken
  - Novartis Investigative Site, Nagano, Nagano
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Kasukabe, Saitama
  - Novartis Investigative Site, Shizuoka, Shizuoka
- Taiwan (3):
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Kaoshiung
  - Novartis Investigative Site, Taipei

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Chen JB, Chiang SS, Chen HC, Obayashi S, Nagasawa M, Hexham JM, Balfour A, Junge G, Akiba T, Fukagawa M. Efficacy and safety of SBR759, a novel calcium-free, iron(III)-based phosphate binder, in Asian patients undergoing hemodialysis: A 12-week, randomized, open-label, dose-titration study versus sevelamer hydrochloride. Nephrology (Carlton). 2011 Nov;16(8):743-50. doi: 10.1111/j.1440-1797.2011.01509.x. PMID 21854503